CLINICAL TRIAL: NCT03164759
Title: Correlation Between Radiographic Bone Density in CBCT and Implant Stability Quotient Value: Clinical Observational Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohammed Basyoni Mohammed Abo El Azem, Principle investigator, Cairo University
Other Study IDs: CEBC-CU-2017-05-23
Record Dates: First submitted 2017-05-22; First posted 2017-05-24 (Actual); Last update posted 2017-05-24 (Actual); Status verified 2017-05

CONDITIONS: Dental Implantation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Correlate the implant stability quotient values measured by ostell device with radiographic bone density measured on CBCT by bluesky software pre-operatively

DETAILED DESCRIPTION:
Dental implants have been widely used in the field of dental rehabilitation. Nowadays implant sucess rate is very high but to keep faliure rate as low as possible patient selection is very important especially regarding bone density to achieve high primary stability. Primary stability plays an important role in successful osteointegration of dental implants. This study was done to correlate between the bone density pre operatively measured on CBCT represented by HF unit and implant stability measured post operatively by ostell device represented by ISQ unit

ELIGIBILITY:
Inclusion Criteria:

* patients receiving dental implants in both arches
* patients should be free from any systemic diseases that may affect normal healing of bone, and predicated outcome
* no intra-oral soft tissue defect that would render primary closure of the intra-oral wound

Exclusion Criteria:

* patients with systemic diseases

  _ patients with ridge augmentation such as ridge expansion, ridge splitting and bone grafting
* patients with sinus lifting done to place implants
* immediate extraction sockets

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients receiving dental implants in healed non grafted sites in both arches
Sampling Method: Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2017-06-01 (Estimated); Primary Completion 2018-06-01 (Estimated); Study Completion 2018-06-01 (Estimated)

PRIMARY OUTCOMES:
Bone density | Baseline
  Measuring bone density on CBCT by bluesky software representing by hounsfield unit pre operatively
Implant stability | Immediate post operative
  Post oprative measurements of implant stability by ostell device (ISQ)